CLINICAL TRIAL: NCT01058226
Title: Reproducibility of Malaria Challenge in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Angela Talley MD, Lead Trials Investigator, Seattle Biomedical Research Institute
Masking: None
Other Study IDs: MC-001
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Experimental malaria challenge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Malaria challenge (wild-type NF54 strain Plasmodium falciparum sporozoites) — Malaria sporozoite challenge with the wild-type NF54 strain of Plasmodium falciparum delivered by the bite of five infected Anopheles stephensi mosquitoes.

SUMMARY:
This is a prospective, single arm, single intervention safety and immunogenicity study in 6 healthy, malaria-naive adults, conducted to demonstrate the successful implementation of the well-established malaria challenge model at the Seattle Biomedical Research Institute (Seattle BioMed).

DETAILED DESCRIPTION:
This study is designed to demonstrate the ability to inoculate malaria naive human volunteers with the Plasmodium falciparum strain of malaria sporozoites by the bite of infected mosquitoes under controlled conditions. Subjects are monitored closely for development of malaria and treated with standard doses of anti-malarial medications which the Plasmodium falciparum strain of malaria is known to be sensitive.

Study participants will undergo malaria sporozoite challenge with wild-type NF54 strain of Plasmodium falciparum sporozoites administered via the bite of five infected Anopheles stephensi mosquitoes under controlled containment conditions.

Participants will be closely monitored for acute reactogenicity and signs and/or symptoms of malaria infection, and from day five post-challenge, will have daily blood films examined for the presence of malaria parasites. Participants who develop malaria infection will be treated with a standard oral regimen of chloroquine, or other FDA-approved anti-malarial drugs, under direct observation. Participants will be treated upon first evidence of microscopic parasitemia or at day 18 if they remain negative. Participants will be housed with study staff in a local hotel for close observation from day 9 post-challenge, until three consecutive blood smears are negative and all symptoms have resolved, then followed weekly for a total of 8 weeks.

Follow-up for safety will be conducted at 4- and 6- months post-challenge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Male or non-pregnant female
* Good general health
* Hemoglobin, WBC, platelets and creatinine within normal ranges
* ALT, AST, bilirubin, alkaline phosphatase <1.25 times upper limit of normal
* Normal urine
* Negative HIV-1 and 2 blood test
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV)
* Low risk for coronary heart disease (CHD)
* Ability and willingness to provide informed consent
* Assessment of Understanding questionnaire completed
* Reliable access to the trial center and availability for duration of study
* If the participant is biologically female, she must:

  * Have negative serum or urine beta human chorionic gonadotropin pregnancy test performed within 3 days prior to challenge
  * Agree to consistently use effective contraception from 21 days prior to enrollment for the duration of the study
  * OR not be of reproductive potential
  * OR be sexually abstinent
  * Also agree not to seek pregnancy through alternative methods

Exclusion Criteria:

* Planned travel to malaria endemic area during the study period
* Recent travel to a malaria endemic area within 3 months of enrollment
* Prior receipt of an investigational malaria vaccine
* History of malaria diagnosis based on positive peripheral blood smear
* Use of malaria chemoprophylaxis with chloroquine within 5 months of malaria challenge, with atovaquone/proguanil within 2 months of malaria challenge or with mefloquine within 30 days prior to malaria challenge
* Recent or anticipated use of systemic antibiotics with anti-malarial effects during the study period
* Anticipated use of medications known to interact with chloroquine and/or atovaquone/proguanil during the study period
* Use of investigational or non-registered drug or vaccine within 30 days preceding challenge or planned use during the study period
* Immunosuppressive medications received within 6 months prior to challenge or planned use within 21 days after challenge
* Any vaccination received or planned within 30 days prior to challenge
* Blood products or immunoglobulins received within 120 days of challenge
* Screening laboratory abnormalities
* Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status
* History of anaphylaxis
* History of severe allergic reactions to mosquito bites
* History of, or known active cardiac disease
* Elevated risk of coronary heart disease
* Clinically significant ECG findings
* Chronic or active neurologic disease
* History of splenectomy or functional asplenia
* History of psoriasis or porphyria
* History of ocular disease diagnosed by an ophthalmologist as retinopathy or visual field defects
* Acute illness at the time of enrollment
* Serologic positivity for HIV, hepatitis C and/or hepatitis b
* Pregnant or lactating female or female who intends to become pregnant during the study period
* Psychiatric condition that precludes compliance with the protocol including but not limited to: psychosis within the past 3 years OR ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV
* Recreational intravenous drug use in the last 12 months
* Any other finding that, in the judgement of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent or increase the risk of having an adverse outcome from participating in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Development of malaria parasitemia and time to parasitemia demonstrated on peripheral blood smear | Day 5 through Day 28 post challenge

SECONDARY OUTCOMES:
Occurrence of unsolicited AEs | Day 0 through Day 56 post challenge
Local and systemic solicited adverse events (AEs) | Day 5 through Day 28 post challenge
Occurrence of serious AEs | Day 0 through Day 56 post challenge
Cell-mediated immune response to experimental malaria infection | Day 0 through Day 56 post challenge
Humoral immune responses to experimental malaria infection | Day 0 through Day 56 post challenge

CONTACTS AND LOCATIONS:
Overall Officials: Angela Talley, M.D., Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Biomedical Research Institue's Malaria Clinical Trial Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Talley AK, Healy SA, Finney OC, Murphy SC, Kublin J, Salas CJ, Lundebjerg S, Gilbert P, Van Voorhis WC, Whisler J, Wang R, Ockenhouse CF, Heppner DG, Kappe SH, Duffy PE. Safety and comparability of controlled human Plasmodium falciparum infection by mosquito bite in malaria-naive subjects at a new facility for sporozoite challenge. PLoS One. 2014 Nov 18;9(11):e109654. doi: 10.1371/journal.pone.0109654. eCollection 2014. PMID 25405724